CLINICAL TRIAL: NCT01405118
Title: A Phase 1, Open Labeled, Fixed Sequence Study To Estimate The Effect Of CP-690,550 On The Pharmacokinetics Of Metformin In Healthy Volunteers
Brief Title: Effect Of CP-690,550 On The Pharmacokinetics Of Metformin In Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: A3921143
Record Dates: First submitted 2011-07-07; First posted 2011-07-29 (Estimated); Last update posted 2011-08-18 (Estimated); Status verified 2011-08

CONDITIONS: Rheumatoid Arthritis
Keywords: Drug-Drug Interaction Healthy Volunteers CP-690; 550 Metformin
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Metformin/CP-690,550 (Experimental)
  Interventions: Drug: Metformin/CP-690,550

INTERVENTIONS:
Drug: Metformin/CP-690,550 — Single oral 500 mg dose of metformin on Days 1 and 4 and multiple oral 30 mg doses of CP-690,550 every 12 hours on Days 2-4.

SUMMARY:
This study will evaluate the potential effect of CP 690,550 on the pharmacokinetics of metformin, a probe drug for organic cationic transport.

ELIGIBILITY:
Inclusion Criteria:

* Adult healthy male and/or female (of non child bearing potential) subjects.

Exclusion Criteria:

* Subjects with clinically significant systemic and laboratory abnormalities.
* Subjects with clinically significant infections within the past 3 months.
* Women of child-bearing potential.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2011-06; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
AUCinf (Area under the plasma concentration-time profile from time zero extrapolated to infinite time) of metformin | 0.5, 1.5, 2, 3, 4, 6, 8, 9, 10, 12 and 24 hours after the metformin dose on Day 4
Cmax (Maximum plasma concentration) of metformin | 0.5, 1.5, 2, 3, 4, 6, 8, 9, 10, 12 and 24 hours after the metformin dose on Day 4
Clr (Renal clearance) of metformin | 0.5, 1.5, 2, 3, 4, 6, 8, 9, 10, 12 and 24 hours after the metformin dose on Day 4

SECONDARY OUTCOMES:
AUClast (Area under the plasma concentration-time profile from time zero to the time of the last quantifiable concentration) of metformin | 0.5, 1.5, 2, 3, 4, 6, 8, 9, 10, 12 and 24 hours after the metformin dose on Day 4
t½ (Terminal half-life) of metformin | 0.5, 1.5, 2, 3, 4, 6, 8, 9, 10, 12 and 24 hours after the metformin dose on Day 4
Tmax (Time for maximum plasma concentration) of metformin | 0.5, 1.5, 2, 3, 4, 6, 8, 9, 10, 12 and 24 hours after the metformin dose on Day 4
Ae24 (Cumulative amount of drug recovered unchanged in urine from time zero to 24 hours postdose) of metformin | 0 hours and intervals 0-3, 3-6, 6-9, 9-12 and 12 24 hours after the metformin dose on Day 4
Ae24% (Percent of dose recovered unchanged in urine from time zero to 24 hours postdose) of metformin | 0 hours and intervals 0-3, 3-6, 6-9, 9-12 and 12 24 hours after the metformin dose on Day 4
Clr (Renal clearance) over each collection interval for metformin | 0 hours and intervals 0-3, 3-6, 6-9, 9-12 and 12 24 hours after the metformin dose on Day 4
CP-690,550 plasma concentration at 2 hours postdose | 2 hrs after first CP-690,550 dose on Day 4

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Brussels, Belgium

REFERENCES:
- [Derived] Klamerus KJ, Alvey C, Li L, Feng B, Wang R, Kaplan I, Shi H, Dowty ME, Krishnaswami S. Evaluation of the potential interaction between tofacitinib and drugs that undergo renal tubular secretion using metformin, an in vivo marker of renal organic cation transporter 2. Clin Pharmacol Drug Dev. 2014 Nov;3(6):499-507. doi: 10.1002/cpdd.120. Epub 2014 May 23. PMID 27129125
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3921143&StudyName=Effect%20Of%20CP-690%2C550%20On%20The%20Pharmacokinetics%20Of%20Metformin%20In%20Healthy%20Volunteers%20